CLINICAL TRIAL: NCT01389232
Title: The SeriScaffold® Use in Reconstruction Post Market Study for Tissue Support and Repair in Breast Reconstruction Surgery in Europe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURE-002
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Soft Tissue Support and Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SeriScaffold® Surgical Scaffold (Experimental): Participants with breast reconstruction surgery implanted with SERI® Surgical Scaffold.
  Interventions: Device: SeriScaffold® Surgical Scaffold

INTERVENTIONS:
Device: SeriScaffold® Surgical Scaffold — A CE Marked, 510(k) cleared, knitted, multi-filament, bioengineered, silk mesh indicated for use as a transitory scaffold for soft tissue support and repair

SUMMARY:
This is a post-market study of the use of SeriScaffold® for soft tissue support and repair in breast reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be female, greater or equal to 18 years of age
* Be willing to undergo immediate breast reconstruction with sub-pectoralis muscle placement of a breast implant
* Be willing to undergo mastectomy with healthy, well vascularized skin flaps anticipated by the surgeon
* Be in good health other than breast pathology and be suited to general anesthesia and planned treatments

Exclusion Criteria:

* Have undergone breast radiation treatment and/or is preoperatively evaluated to require radiation treatment to the breast area during the course of the study
* Have a known allergy to silk
* Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability
* Have undergone previous breast surgery with the exception of mastectomy, breast biopsy, cyst removal, lumpectomy, mastopexy, reduction and/or augmentation
* Have had a prior soft tissue support device implanted in the breast
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (2):
  - Düsseldorf
  - Munich
- Milan, Italy
- Barcelona, Spain
- Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was defined as having signed the IRB-approved Informed Consent Form. 104 participants were enrolled, of which 100 were implanted with SERI® Surgical Scaffold and are presented in the participant flow.
Period: Overall Study
Arm/Group | SeriScaffold® Surgical Scaffold
Started | 100
Completed | 81
Not Completed | 19
Not completed — Had scaffold removed | 15
Not completed — Personal reasons | 2
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Subjects implanted with SERI® during their Stage I breast reconstruction surgery
Arm/Group | SeriScaffold® Surgical Scaffold
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator Satisfaction With Seri® Surgical Scaffold on an 11-Point Scale
Description: Investigator satisfaction after stage I surgery/implantation of SERI® Surgical Scaffold is evaluated on an 11-point scale, where 0=very dissatisfied to 10=very satisfied.
Time Frame: Month 6
Population: All participants with a Month 6 visit. 12 subjects exited the study prior to Month 6.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | SeriScaffold® Surgical Scaffold
Number analyzed (Participants) | 88
Scores on a Scale | 8.8 (1.5)

2. Secondary Outcome: Investigator Satisfaction With Seri® Surgical Scaffold on an 11-Point Scale
Description: as for outcome 1
Time Frame: Month 3, Month 12, Month 18, Month 24
Population: All participants with a visit at the designated time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | SeriScaffold® Surgical Scaffold
Number analyzed (Participants) | 89
Scores on a Scale
  Month 3 (N=89) | 8.6 (1.5)
  Month 12 (N=83): number analyzed (Participants) | 83
  Month 12 (N=83) | 8.8 (1.3)
  Month 18 (N=79): number analyzed (Participants) | 79
  Month 18 (N=79) | 8.8 (1.5)
  Month 24 (N=80): number analyzed (Participants) | 80
  Month 24 (N=80) | 9.0 (1.1)

3. Secondary Outcome: Investigator Assessment of Ease of Use of Seri® Surgical Scaffold on a 5-Point Scale
Description: Investigator assessment of ease of use of SERI® Surgical Scaffold is evaluated on a 5-point scale, where 1=very difficult to use to 5=very easy to use.
Time Frame: Immediately Following Stage 1 Surgery
Population: All implanted participants. "Scaffold cutting and sharping before implantation" was reported "Not done" on n=50
Measure: Number; unit: Participants
Groups:
- Ease of Use During Surgery = Very Difficult to Use; Ease of Use During Surgery = Difficult to Use; Ease of Use During Surgery = Neither Difficult Nor Easy to Use; Ease of Use During Surgery = Easy to Use; Ease of Use During Surgery = Very Easy to Use: Implanted Participants: Participants with breast reconstruction surgery implanted with SERI® Surgical Scaffold.
- Not Done: Implanted participants on whom procedure was reported "not done"
Arm/Group | Ease of Use During Surgery = Very Difficult to Use | Ease of Use During Surgery = Difficult to Use | Ease of Use During Surgery = Neither Difficult Nor Easy to Use | Ease of Use During Surgery = Easy to Use | Ease of Use During Surgery = Very Easy to Use | Not Done
Number analyzed (Participants) | 100 | 100 | 100 | 100 | 100 | 100
Participants
  Scaffold preparation before implantation | 0 | 0 | 3 | 20 | 77 | 0
  Scaffold cutting and shaping before implantation | 0 | 1 | 5 | 6 | 38 | 50
  Scaffold positioning/drapability during implant | 0 | 0 | 37 | 14 | 49 | 0
  Scaffold cutting and shaping after implantation | 0 | 1 | 35 | 12 | 52 | 0
  Scaffold suturing during implantation | 0 | 1 | 37 | 14 | 48 | 0

4. Secondary Outcome: Breast Anatomy Measurements
Description: Breast anatomy measurements were taken at the following points: sternal notch to apex, sternal notch to inframammary fold, apex to inframammary fold, and medial mammary fold to lateral mammary fold.
Time Frame: Preoperative, First Postoperative, Month 3, Month 6, Month 12, Month 18, Month 24
Population: All implanted breasts evaluated at the designated time point
Measure: Mean (95% Confidence Interval); unit: Centimeters (cm)
Units Other Than Participants: Breasts
Groups:
- Sternal Notch to Apex; Sternal Notch to Inframammary Fold; Apex to Inframammary Fold; Medial Mammary Fold to Lateral Mammary Fold: Implanted Participants: Participants with breast reconstruction surgery implanted with SERI® Surgical Scaffold.
Arm/Group | Sternal Notch to Apex | Sternal Notch to Inframammary Fold | Apex to Inframammary Fold | Medial Mammary Fold to Lateral Mammary Fold
Number analyzed (Participants) | 100 | 100 | 100 | 100
Number analyzed (Breasts) | 149 | 149 | 149 | 149
Centimeters (cm)
  Preoperative: number analyzed (Participants) | 87 | 87 | 87 | 87
  Preoperative: number analyzed (Breasts) | 132 | 132 | 132 | 132
  Preoperative | 21.3 [20.9 to 21.7] | 24.1 [23.7 to 24.4] | 7.1 [6.9 to 7.2] | 14.6 [14.3 to 14.9]
  First Postoperative: number analyzed (Participants) | 88 | 88 | 88 | 88
  First Postoperative: number analyzed (Breasts) | 133 | 133 | 133 | 133
  First Postoperative | 19.0 [18.7 to 19.2] | 22.6 [22.3 to 22.8] | 8.1 [7.9 to 8.2] | 14.5 [14.3 to 14.8]
  Month 3: number analyzed (Participants) | 87 | 87 | 87 | 87
  Month 3: number analyzed (Breasts) | 130 | 130 | 130 | 130
  Month 3 | 19.0 [18.8 to 19.3] | 22.7 [22.4 to 23.0] | 8.1 [7.9 to 8.3] | 14.2 [14.0 to 14.4]
  Month 6: number analyzed (Participants) | 83 | 83 | 83 | 83
  Month 6: number analyzed (Breasts) | 126 | 126 | 126 | 126
  Month 6 | 19.2 [18.9 to 19.5] | 23.0 [22.7 to 23.2] | 8.1 [7.9 to 8.3] | 14.1 [13.8 to 14.3]
  Month 12: number analyzed (Participants) | 79 | 79 | 79 | 79
  Month 12: number analyzed (Breasts) | 118 | 118 | 118 | 118
  Month 12 | 19.2 [18.9 to 19.4] | 23.0 [22.7 to 23.3] | 8.0 [7.8 to 8.1] | 14.0 [13.7 to 14.3]
  Month 18: number analyzed (Participants) | 69 | 69 | 69 | 69
  Month 18: number analyzed (Breasts) | 101 | 101 | 101 | 101
  Month 18 | 19.0 [18.7 to 19.3] | 22.9 [22.5 to 23.2] | 8.0 [7.8 to 8.1] | 13.7 [13.5 to 14.0]
  Month 24: number analyzed (Participants) | 73 | 73 | 73 | 73
  Month 24: number analyzed (Breasts) | 112 | 112 | 112 | 112
  Month 24 | 19.0 [18.7 to 19.3] | 22.9 [22.6 to 23.2] | 8.1 [7.9 to 8.3] | 13.8 [13.5 to 14.0]

5. Secondary Outcome: Subject Satisfaction With Breasts on a 5-Point Scale
Description: Subject satisfaction with breasts is evaluated on a 5-point scale, where 1=very dissatisfied to 5=very satisfied.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: All implanted breasts evaluated at the designated time point. Data was not available for 1 subject (both breasts) at baseline, 1 subject (right breast) at Month 6, 2 subjects (right breast) at Month 18 and 1 subject (right breast) at Month 24.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Units Other Than Participants: Breasts
Arm/Group | SeriScaffold® Surgical Scaffold
Number analyzed (Participants) | 100
Number analyzed (Breasts) | 146
Scores on a Scale
  Baseline (Missing=0) | 3.7 (1.0)
  Month 6 (Missing=0): number analyzed (Participants) | 88
  Month 6 (Missing=0): number analyzed (Breasts) | 129
  Month 6 (Missing=0) | 4.3 (0.9)
  Month 12 (Missing=1): number analyzed (Participants) | 85
  Month 12 (Missing=1): number analyzed (Breasts) | 125
  Month 12 (Missing=1) | 4.4 (0.8)
  Month 18 (Missing=2): number analyzed (Participants) | 83
  Month 18 (Missing=2): number analyzed (Breasts) | 119
  Month 18 (Missing=2) | 4.4 (0.7)
  Month 24 (Missing=0): number analyzed (Participants) | 81
  Month 24 (Missing=0): number analyzed (Breasts) | 122
  Month 24 (Missing=0) | 4.4 (0.7)

ADVERSE EVENTS:
Description: Subjects implanted with SERI® during their Stage I breast reconstruction surgery were used to evaluate serious adverse events and adverse events.
Arm/Group | SeriScaffold® Surgical Scaffold
Serious Adverse Events (participants affected / at risk) | 53/100
Other Adverse Events (participants affected / at risk) | 92/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SeriScaffold® Surgical Scaffold (N=100)
Neutropenia (Blood and lymphatic system disorders) | 2
Capsular contracture associated with breast implant (General disorders) | 2
Device extrusion (General disorders) | 5
Pyrexia (General disorders) | 3
Mastitis (Infections and infestations) | 2
Neutropenic sepsis (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Seroma (Injury, poisoning and procedural complications) | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 2
Physical examination abnormal (Investigations) | 3
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 6
Haematoma (Vascular disorders) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Device Dislocation (General disorders) | 1
Inflammation (General disorders) | 1
Medical Device Complication (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Endometritis (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Fractured Sacrum (Injury, poisoning and procedural complications) | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Placenta Previa (Pregnancy, puerperium and perinatal conditions) | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SeriScaffold® Surgical Scaffold (N=100)
Capsular contracture associated with breast implant (General disorders) | 7
Device dislocation (General disorders) | 5
Device extrusion (General disorders) | 9
Impaired healing (General disorders) | 5
Implant site reaction (General disorders) | 6
Pyrexia (General disorders) | 9
Gastroenteritis (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 14
Seroma (Injury, poisoning and procedural complications) | 30
Wound dehiscence (Injury, poisoning and procedural complications) | 9
Physical examination abnormal (Investigations) | 8
Headache (Nervous system disorders) | 12
Breast pain (Reproductive system and breast disorders) | 14
Erythema (Skin and subcutaneous tissue disorders) | 18
Skin necrosis (Skin and subcutaneous tissue disorders) | 21
Haematoma (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.